CLINICAL TRIAL: NCT04974073
Title: Development of PHY606 as Adjunct Therapy for Anemia Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sheng-Teng Huang (Other)
Responsible Party: Sponsor-Investigator, Sheng-Teng Huang, Attending Physician, China Medical University Hospital
Organization: China Medical University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: CMUH106-REC3-028
Record Dates: First submitted 2021-07-01; First posted 2021-07-23 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Anemia; Herbal Interaction
Keywords: Anemia; Danggui Buxue Tang; PHY606; Side effects; TCM
MeSH Terms: conditions — Anemia | interventions — danggui buxue decoction

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- control group (No Intervention): with traditional western medicine treatment based on underlined disease
- PHY606 (Experimental): PHY606 7.5gm BID for 3 months
  Interventions: Drug: PHY606
- Healthy group (Other): PHY606 7.5gm BID for 2 days
  Interventions: Drug: PHY606

INTERVENTIONS:
Drug: PHY606 — Danggui Buxue Tang is a well-known TCM formula indicated for anemia through immune modulation and increase energy metabolism
  Other Names: Danggui Buxue Tang
  Arms: Healthy group; PHY606

SUMMARY:
Many reasons can cause anemia, decreased RBC production or increased destruction of circulation RBC. The investigators investigate the Danggui Buxue Tang (PHY606) composed of Angelicae Sinensis Radix and Astragali Radix in the fields of genomic and metabolomics in the healthy people and the patiens with anemia.

DETAILED DESCRIPTION:
Many reasons can cause anemia, decreased RBC production or increased destruction of circulating RBC. The reasons of the former are lake of nutrients, bone marrow disorder, low level tropic hormone, inflammation associated with infectious, inflammatory, or malignant disorders and the latter are intravascular hemolysis or blood loss. Anemia is characterized by the sign of pallor (reduced oxyhemoglobin in skin or mucous membranes), fatigue, lightheadedness, and weakness associated with low hemoglobin.

Iron deficiency anemia (IDA) is mainly resulted from inadequate iron uptake of food, malabsorption of iron and blood loss. Adult female are easy to have IDA compared to male because of menstruation, pregnancy, lactation and low caloric uptake leading to iron deficiency. In Taiwan, cancer-related and chronic kidney disease also lead to insufficient secretion of erythropoietin (EPO). The cost of long-term use EPO and its derivative drugs is high. Besides, drug resistance, risk of tumor growth and cardiovascular disease are all important issues. However, ferrotherapy will induce GI upset, muscle pain and skin hives. Also, iron supplementation can lead to an increase in infectious disease morbidity in areas where bacterial infections or where malaria are common.

Based on the concept of dietetic invigoration, the investigators investigate the Danggui Buxue Tang (PHY606) composed of Angelicae Sinensis Radix and Astragali Radix in the fields of genomics and metabolomics in the healthy people and the patients with anemia. In the meantime, the investigators will explore whether PHY606 activates the immune function, improves anemia and reduces the side effects induced by anemia treatment. Furthermore, the novel metabolites from Angelicae Sinensis Radix and Astragali Radix will be tested from clinic back to the bench including immunological potentiation and hematopoietic function. According to the TCM theory, the investigators integrate with modern medicine and molecular biotechnology to investigate anemia and hope to provide the evidence base for clinical application.

ELIGIBILITY:
Inclusion Criteria:

* female: Hb<11 g/dL; male: Hb<13.5 g/dL
* has no allergic reaction to TCM

Exclusion Criteria:

* below 20 years old
* ever drug abuse or still in drug abuse
* pregnant or in breast-feeding women
* with psychotic disorders
* cardiac arrhythmia with pacemaker
* dyscoagulation or thrombocytopenia (platelet< 15000/uL) or liver dysfunction (> 2 fold normal range)
* with severe disease (cardiac arrest, heart failure, COPD, GI bleeding, etc.)
* under another clinical trials

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2017-08-22 (Actual); Primary Completion 2017-08-22 (Actual); Study Completion 2019-11-18 (Actual)

PRIMARY OUTCOMES:
Constitution in Chinese Medicine Questionnaire (CCMQ) | Change from baseline CCMQ at Day0, Day31, Day93 and Day180.
Serum Cytokines | Change from baseline serum cytokines at Day0, Day31 and Day93.
  Collect blood and measure the level of serum cytokines.

SECONDARY OUTCOMES:
Tongue diagnosis | Change from baseline tongue diagnosis at Day0 and Day93.
  Use tongue photos for analysis
Pulse diagnosis | Change from baseline Pulse diagnosis at Day0 and Day93.
  Use the pulse detector to detect the rhythm data of the subject's left and right hand pulse.
Anemia blood test | Change from baseline anemia blood at Day 0, Day 31 and Day93.
  Collect blood and measure the level of ferritin(ng/mL), TIBC(ug/dL), transferrin(mg/dL).
Genotype | Change from baseline genotype at Day 0, Day 31 and Day93.
  Collect blood and analyze the genotype by microarray assay.

OTHER OUTCOMES:
Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) | Change from baseline FACIT-F score at Day0, Day31, Day93 and Day180.
Pittsburgh Sleep Quality Index (PSQI) | Change from baseline PSQI score at Day0, Day31, Day93 and Day180.
36-Item Short Form Health Survey (SF-36) | Change from baseline SF-36 score at Day0, Day31, Day93 and Day180.
White blood cell (WBC) | Change from baseline WBC at Day 0, Day 31 and Day93.
  Collect blood and measure the value of WBC (x 10^3/ul).
Red Blood Cells (RBC) | Change from baseline RBC at Day 0, Day 31 and Day93.
  Collect blood and measure the value of RBC (x 10^6/ul).
Hemoglobin (Hb) | Change from baseline Hemoglobin at Day 0, Day 31 and Day93.
  Collect blood and measure the value of Hemoglobin (gm/dL).
Hematocrit (Hct) | Change from baseline Hematocrit at Day 0, Day 31 and Day93.
  Collect blood and measure the value of Hematocrit (%).
Red blood cell volume distribution width (RDW) | Change from baseline RDW at Day 0, Day 31 and Day93.
  Collect blood and measure the value of RDW (%).
Platelet | Change from baseline Platelet at Day 0, Day 31 and Day93.
  Collect blood and measure the value of Platelet (x 10^3/ul).
Mean corpuscular volume (MCV) | Change from baseline MCV at Day 0, Day 31 and Day93.
  Collect blood and measure the value of MCV (fl).
Mean corpuscular hemoglobin (MCH) | Change from baseline MCH at Day 0, Day 31 and Day93.
  Collect blood and measure the value of MCH (pg).
Mean corpuscular hemoglobin concentration (MCHC) | Change from baseline MCHC at Day 0, Day 31 and Day93.
  Collect blood and measure the value of MCHC (g/dL).
Mean platelet volume (MPV) | Change from baseline MPV at Day 0, Day 31 and Day93.
  Collect blood and measure the value of MPV (fl).

CONTACTS AND LOCATIONS:
Overall Officials: Sheng-Teng Huang, MD PHD, Principal Investigator — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided